CLINICAL TRIAL: NCT05056532
Title: Evaluation of Primary and Accessory Respiratory Muscles and Their Influence on Exercise Capacity and Dyspnea in Pulmonary Arterial Hypertension
Brief Title: Evaluation of Respiratory Muscle in Patient With Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Other Study IDs: PAH
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Artery Hypertension
Keywords: respiratory muscle strength; exercise capacity; dyspnea; accessory respiratory muscle
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: Maximal mouth pressure will be evaluated for determine respiratory muscle strength, m. pectoralis, m. serratus anterior, m. sternocloideumasteoideus and quadriceps muscles strengths will be measured to evaluate accessory respiratory muscle strength, London chest activity of daily living scale will be done for assessment of dyspnea and six minute walk test will be used for determination of functionally capacity
  Interventions: Diagnostic Test: patient assessment
- Control group: Maximal mouth pressure will be evaluated for determine respiratory muscle strength, m. pectoralis, m. serratus anterior, m. sternocloideumasteoideus and quadriceps muscles strengths will be measured to evaluate accessory respiratory muscle strength, London chest activity of daily living scale will be done for assessment of dyspnea and six minute walk test will be used for determination of functionally capacity
  Interventions: Diagnostic Test: patient assessment

INTERVENTIONS:
Diagnostic Test: patient assessment — subjective and objective measurement will be performed in patients with PAH

SUMMARY:
The aim of the study is that evaluation of basic and accessory respiratory muscles and their relationship of six minute walk test in patient with pulmonary arterial hypertension (PAH)

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of pulmonary arterial hypertension
* patients with stabil drug therapy at least three months

Exclusion Criteria:

* patients with obstructive and/ or restrictive lung disease comorbidity
* severe orthopedic and/ or neurological comorbidity
* patients with heart failure
* patients with ischemic heart disease
* uncooperative patients

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patient group will be chosen among the admitted to clinic control group will consist of invited volunteers
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
pectoralis muscle strength | 15 minute
  pectoralis muscle strength will be evaluated with hand held dynamometers according to muscle test technique
serratus anterior muscle strength | 15 minutes
  Serratus anterior muscle strength will be evaluated with hand held dynamometers according to muscle test technique
sternocleidomasteoideus muscle strength | 15 minutes
  sternocleidomasteoideus muscle strength will be evaluated with hand held dynamometers according to muscle test technique
Respiratory mouth pressure | 15 minutes
  Respiratory mouth pressure will be measured to determine maximally inspiratory pressure and maximally expiratory pressure according to ATS/ERS guidelines.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) | 30 minutes
  Six minute walk test will be performed to evalute functionally exercise capacity according to ATS/ERS guidelines
Dyspnea assessment | 20 minutes
  London Chest Activity of Daily Living Scale will be used to sensation of dyspnea during activity of daily living.The scale consists of four domains: self-care (four items), domestic (six items), physical (two items) and leisure (three items). In total, the scale consisting of 15 items scored of 0 to 5. 0 means that "I wouldn't do anyway" and 5 means that "Someone else does it for me". Higher values indicate greater limitation due to the dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Habibe DURDU, Principal Investigator — Giresun University
Locations (1):
- Istanbul university-cerrahpasa cardiology institute, Istanbul, Haseki, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panagiotou M, Peacock AJ, Johnson MK. Respiratory and limb muscle dysfunction in pulmonary arterial hypertension: a role for exercise training? Pulm Circ. 2015 Sep;5(3):424-34. doi: 10.1086/682431. PMID 26401245
- [Background] Riou M, Pizzimenti M, Enache I, Charloux A, Canuet M, Andres E, Talha S, Meyer A, Geny B. Skeletal and Respiratory Muscle Dysfunctions in Pulmonary Arterial Hypertension. J Clin Med. 2020 Feb 3;9(2):410. doi: 10.3390/jcm9020410. PMID 32028638